CLINICAL TRIAL: NCT03739853
Title: Clinical Effectiveness of Standard Step up Care (Methotrexate) Compared to Early Combination DMARD Therapy With Standard Step up Care Compared to Early Use of TNF Inhibitors With Standard Step up Care for the Treatment of Moderate to Severe Psoriatic Arthritis: a 3-arm Parallel Group Randomised Controlled Trial.
Brief Title: Severe Psoriatic Arthritis - Early intervEntion to Control Disease: the SPEED Trial
Acronym: SPEED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 18/SC/0107
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-12

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Methotrexate; Sulfasalazine; Leflunomide; Adalimumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded assessor will perform clinical evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard care (Active Comparator): Control 'step-up' therapy in the cohort (MONITOR-PsA study). Therapy for the cohort is defined by standard NHS practice following international recommendations and National requirements for the prescription of biologic therapy[19-22]. Commonly Initial therapy will be with methotrexate alone (15mg/week rising to 25mg/week as tolerated by week 8 of therapy) unless this is contraindicated. In cases of non-response or intolerance to methotrexate, participants will have an alternative DMARD (most commonly sulfasalazine or leflunomide) added or switched to. In cases of failure of two DMARDs, treatment can be escalated to biologic therapy as per National Institute for Health and Clinical Excellence (NICE) recommendations. If the requisite disease activity is not met or if there are contraindications to biologics, alternative DMARD combinations will be used.
  Interventions: Drug: Methotrexate; Drug: Sulfasalazine; Drug: Leflunomide
- Combination csDMARD (Experimental): Arm 2 - Combination DMARD arm. All participants will be prescribed methotrexate with an additional DMARD (either sulfasalazine or leflunomide) at baseline. Response will be assessed after 12 weeks of therapy using the Minimal Disease Activity (MDA) criteria. Participants who achieve the MDA criteria by week 12 on this combination therapy will continue . Participants who show a significant response by in week 12 (a reduction in tender and swollen joint counts of at least 20%) but do not yet meet the MDA criteria should continue on this therapy for an additional 12 weeks before review. Participants failing to show significant response (reduction in joint counts by less than 20%) by week 12 on this combination therapy or those failing to meet MDA criteria by week 24 will be eligible for rescue therapy
  Interventions: Drug: Methotrexate; Drug: Sulfasalazine; Drug: Leflunomide
- Early TNF inhibition (Experimental): Early biologic arm. All participants will be prescribed methotrexate (given weekly) with a TNF inhibitor (adalimumab given every two weeks) at baseline. Treatment with TNF inhibitor will be continued until week 24 at which time the TNF inhibitor will be tapered to week 32. The TNF inhibitor will be stopped completely after week 32 and participants will continue on methotrexate. In case of flare of disease, participants will be eligible for rescue therapy
  Interventions: Drug: Methotrexate; Drug: Adalimumab

INTERVENTIONS:
Drug: Methotrexate — Used in all three arms of study
Drug: Sulfasalazine — Used in arm 2 of study
  Arms: Combination csDMARD; Standard care
Drug: Leflunomide — Used in arm 2 of study
  Arms: Combination csDMARD; Standard care
Drug: Adalimumab — Used in arm 3 of the study only
  Arms: Early TNF inhibition

SUMMARY:
SPEED is a three arm interventional trial nested within a cohort (Trials Within Cohorts or TWiCs design). This tests more aggressive early therapy in patients newly diagnosed with moderate to severe PsA. Arm 1 will receive standard step up therapy in the cohort and act as the control group. Arm 2 will receive early combination conventional synthetic disease modifying anti-rheumatic drugs (csDMARDs). Arm 3 will receive early tumour necrosis factor (TNF) inhibitor therapy.

DETAILED DESCRIPTION:
Arm 1: Control 'step-up' therapy in the cohort (MONITOR-PsA study). Therapy for the cohort is defined by standard practice in these PsA clinics following current international recommendations[11] and National requirements for the prescription of biologic therapy[19-22]. Whilst physician discretion is used, most commonly Initial therapy will be with methotrexate alone (15mg/week rising to 25mg/week as tolerated by week 8 of therapy) unless this is contraindicated. In cases of non-response or intolerance to methotrexate, participants will have an alternative DMARD (most commonly sulfasalazine or leflunomide) added or switched to at the discretion of the rheumatologist. In cases of failure of two DMARDs, treatment can be escalated to biologic therapy as per National Institute for Health and Clinical Excellence (NICE) recommendations[19-22] usually with a TNF inhibitor as first line. If the requisite disease activity is not met or if there are contraindications to biologics, alternative DMARD combinations will be used. Further details are available in the PsA clinic treatment protocol which is Appendix D in the MONITOR-PsA protocol.

ARM 2: Combination DMARD arm. All participants will be prescribed methotrexate with an additional DMARD (either sulfasalazine or leflunomide) at baseline, staggering the start of these additional therapies by one week to allow more accurate attribution of adverse events. Either sulfasalazine or leflumonide will be used in combination depending on physician preference (taking into account disease presentation, arthritis, enthesitis, skin disease, risk of hypertension and liver disease).Response will be assessed after 12 weeks of therapy using the Minimal Disease Activity (MDA) criteria. These assess 7 different outcomes and patients should meet at least 5 of the 7 items to be classified as being in MDA. Participants who achieve the MDA criteria by week 12 on this combination therapy will continue on this therapy. Participants who show a significant response by in week 12 (a reduction in tender and swollen joint counts of at least 20%) but do not yet meet the MDA criteria should continue on this therapy for an additional 12 weeks before review. Participants failing to show significant response (reduction in joint counts by less than 20%) by week 12 on this combination therapy or those failing to meet MDA criteria by week 24 will be eligible for rescue therapy following the standard PsA clinic treatment protocol (as per arm 1 above and as detailed in the PsA clinic treatment protocol which is found in appendix D of the MONITOR-PsA protocol). Participants may be eligible at this time point for biologic therapy most commonly using TNF inhibitors under NICE guidelines. These state that patients should have failed adequate trials of at least 2 standard DMARDs and that they should have active disease defined as at least 3 tender and 3 swollen joints. If they do not fulfil these NICE criteria (≥3 tender and ≥3 swollen joints) they will be prescribed alternative DMARDs.

ARM 3: Early biologic arm. All participants will be prescribed methotrexate (given weekly) with a TNF inhibitor (adalimumab given every two weeks) at baseline staggering the start of these therapies by one week to allow more accurate attribution of adverse events (TNF inhibitor from week 0, methotrexate from week 1). Treatment with TNF inhibitor will be continued until week 24 at which time the TNF inhibitor will be tapered by spacing out doses which will be received at week 28 and week 32. The TNF inhibitor will be stopped completely after week 32 and participants will continue on methotrexate. In case of flare of disease, participants will be eligible for rescue therapy following the standard PsA clinic treatment protocol (as per arm 1 above and as detailed in the PsA clinic treatment protocol which is found in appendix D of the MONITOR-PsA protocol). According to this protocol they will be started on combination DMARD therapy (sulfasalazine or leflunomide) and may subsequently be eligible for further TNF inhibitor treatment at a later point if they fulfil NICE criteria (as above).

The Investigational Medicinal Products (IMPs) used in this trial are methotrexate, sulfasalazine, leflunomide and adalimumab. All of these medications are used routinely in PsA patients in standard care.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 18 years or above.
* Participants consented to the PsA inception cohort (MONITOR-PsA) and to be approached for alternate interventional therapies.
* Poor prognostic factors at baseline. Either

  * Polyarticular disease with ≥5 active joints at baseline assessment OR
  * Oligoarticular disease with <5 active joints at baseline but with one or more of the following poor prognostic factors: raised C reactive protein, radiographic damage, health assessment questionnaire>1
* Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the trial and for 3 months thereafter (or 2 years if received leflunomide unless treated with washout therapy) as in standard practice.
* Participant has clinically acceptable laboratory results within 28 days of baseline:

  * Haemoglobin count > 8.5 g/dL
  * White blood count (WBC) > 3.5 x 109/L
  * Absolute neutrophil count (ANC) > 1.5 x 109/L
  * Platelet count > 100 x 109/L
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) and alkaline phosphatase levels <3 x upper limit of normal
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Willing to allow his or her general practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* Previous treatment for articular disease with DMARDs including, but not limited to, methotrexate, sulfasalazine, leflunomide and ciclosporin
* Female patient who is pregnant, breast-feeding or planning pregnancy during the course of the trial.
* Significant renal (estimated glomerular filtration rate <30ml/min) or hepatic impairment.
* Patients who test positive for Hepatitis B, C or HIV.
* Contraindication to any of the investigative drugs.
* Patients who currently abuse drugs or alcohol
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Patient with life expectancy of less than 6 months.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put patients at risk because of participation in the trial, or may influence the result of the trial, or their ability to participate in the trial.
* Participation in another research trial involving an investigational product in the past 12 weeks.

Additional exclusion criteria apply to patients randomised to arm 3 and receiving adalimumab therapy:

* Active tuberculosis (TB), chronic viral infections, recent serious bacterial infections, those receiving live vaccinations within 3 months of the anticipated first dose of study medication, or those with chronic illnesses that would, in the opinion of the investigator, put the participant at risk.
* Latent TB unless they have received appropriate anti-tuberculous treatment as per local guidelines
* History of cancer in the last 5 years, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watson M, Tillett W, Jadon D, Massa MS, Francis A, Gullick N, Rombach I, Sinomati Y, Tucker L, Coates LC. The protocol of a clinical effectiveness trial comparing standard step-up care, early combination DMARD therapy and early use of TNF inhibitors for the treatment of moderate to severe psoriatic arthritis: the 3-arm parallel group SPEED randomized controlled trial. Ther Adv Musculoskelet Dis. 2024 May 30;16:1759720X241240913. doi: 10.1177/1759720X241240913. eCollection 2024. PMID 38826570

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Combination csDMARD | Early TNF Inhibition
Started | 64 | 63 | 65
Completed | 58 | 60 | 62
Not Completed | 6 | 3 | 3

BASELINE CHARACTERISTICS:
Population: No difference
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Combination csDMARD | Early TNF Inhibition | Total
Number analyzed (Participants) | 64 | 63 | 65 | 192
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [34 to 57] | 51 [37 to 60] | 48 [34 to 57] | 49 [34 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 28 | 92
  Male | 33 | 30 | 37 | 100
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 64 | 63 | 65 | 192

OUTCOME MEASURES:

1. Primary Outcome: Psoriatic Arthritis Disease Activity Score (PASDAS)
Description: A composite measure of PsA disease activity. This score is a composite measure of disease activity in PsA. There is only one total score which ranges from 0-10 with higher numbers indicating more active disease. Low disease activity is defined as <3.2.
Time Frame: 24 weeks
Population: With complete data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Combination csDMARD | Early TNF Inhibition
Number analyzed (Participants) | 39 | 47 | 53
score on a scale | 4.7 (1.5) | 4.0 (1.5) | 3.6 (1.9)

2. Secondary Outcome: Psoriatic Arthritis Disease Activity Score (PASDAS)
Description: as for outcome 1
Time Frame: 48 weeks
Population: with complete data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Combination csDMARD | Early TNF Inhibition
Number analyzed (Participants) | 45 | 45 | 49
score on a scale | 4.1 (1.8) | 3.8 (1.5) | 3.5 (1.7)

3. Secondary Outcome: Minimal Disease Activity (MDA)
Description: Response will be assessed after 12 weeks of therapy using the Minimal Disease Activity (MDA) criteria. These assess 7 different outcomes and patients should meet at least 5 of the 7 items to be classified as being in MDA. The MDA criteria are shown in the box below:
  Outcome Measure (see Section 8) Score +1 for each outcome measure which is below the value below.
  Total score of ≥5 indicates MDA achieved Tender joint count (TJC) (using 68 joint count) ≤1 Swollen joint count (SJC) (using 66 joint count) ≤1 Enthesitis count (using LEI or SPARCC) ≤1 Skin assessment PASI≤1 or BSA≤3% Patient global VAS (mm) ≤20 Patient pain VAS (mm) ≤15 HAQ ≤0.5
Time Frame: 12, 24, 36, 48 weeks
Population: Enrolled in study
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Combination csDMARD | Early TNF Inhibition
Number analyzed (Participants) | 64 | 63 | 65
Participants
  Week 12 | 44 | 40 | 42
  Week 24: number analyzed (Participants) | 42 | 51 | 54
  Week 24 | 38 | 36 | 36
  Week 36: number analyzed (Participants) | 38 | 38 | 48
  Week 36 | 30 | 23 | 30
  Week 48: number analyzed (Participants) | 44 | 45 | 51
  Week 48 | 33 | 33 | 35

4. Secondary Outcome: Psoriatic Arthritis Impact of Disease (PsAID)
Description: A questionnaire assessing the overall impact of disease on a patient. This is a scale of 12 questions (scored 0-10) which are combined with published weighting scales to one final 0-10 score where 0 is "no impact" and 10 is "maximal impact". There are no subscales. Patient acceptable symptom state is <=4.
Time Frame: 12, 24, 36, 48 weeks
Population: ITT
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Standard Care | Combination csDMARD | Early TNF Inhibition
Number analyzed (Participants) | 64 | 63 | 65
score on a scale
  Week 12 | 3.9 (2.2) | 4.4 (2.7) | 3.5 (2.3)
  Week 24 | 3.8 (2.1) | 3.5 (2.4) | 3.1 (2.5)
  Week 36 | 3.2 (2.1) | 2.9 (2.4) | 3.3 (2.3)
  Week 48 | 3.4 (2.5) | 3.3 (2.6) | 3.0 (2.5)

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Standard Care | Combination csDMARD | Early TNF Inhibition
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63 | 0/65
Serious Adverse Events (participants affected / at risk) | 2/64 | 0/63 | 2/65
Other Adverse Events (participants affected / at risk) | 19/64 | 20/63 | 18/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=64) | Combination csDMARD (N=63) | Early TNF Inhibition (N=65)
Cerebrovascualr haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Cerebrovascualr haemorrhage confirmed on brain imaging. No sequelae
perineal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Perineal abscess requiring drain and antibiotics
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Admitted briefly for treatment of gastroenteritis.
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Admitted for antibiotics
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=64) | Combination csDMARD (N=63) | Early TNF Inhibition (N=65)
Headache (Nervous system disorders) | 9 (9) | 11 (11) | 5 (5) — Headache
Nausea (Gastrointestinal disorders) | 19 (19) | 20 (20) | 15 (15) — Nausea
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 8 (8) | 6 (6) — Diarrhoea
Liver function test abnormalities (Hepatobiliary disorders) | 11 (11) | 19 (19) | 18 (18) — LFTs above normal range
Infection (Infections and infestations) | 3 (3) | 3 (3) | 6 (6) — Any infection

LIMITATIONS AND CAVEATS:
Some missing data in primary and secondary outcomes due to COVID and other missed visits

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT03739853/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT03739853/SAP_001.pdf